CLINICAL TRIAL: NCT03187223
Title: A Randomized Phase II Trial Comparing Bendamustine and Melphalan With Melphalan Alone as Conditioning Regimen for Autologous Stem Cell Transplantation (ASCT) in Myeloma Patients
Brief Title: Bendamustine and Melphalan in Myeloma
Acronym: BEB-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Mundipharma Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEB-2 Trial
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bendamustine; Melphalan; ASCT
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Bendamustine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Randomized prospective non-blinded clinical phase II trial investigating the drugs bendamustine hydrochloride and melphalan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Mel) (Active Comparator): Melphalan 100mg/m2/day iv days -2 and -1
  Interventions: Drug: Melphalan
- Arm B (BenMel) (Experimental): Melphalan 100mg/m2/day iv days -2 and -1 Bendamustine 200mg/m2/day iv days -4 and -3
  Interventions: Drug: Melphalan; Drug: Bendamustine

INTERVENTIONS:
Drug: Melphalan — High-dose chemotherapy regimen for conditioning treatment before autologous stem cell Transplantation. Patients will receive melphalan at a total dose of 200mg/m2, divided in two doses of 100mg/m2/day on days -2 and -1, with the ASCT at day 0.
  Other Names: Alkeran
Drug: Bendamustine — High-dose chemotherapy regimen for conditioning treatment before autologous stem cell Transplantation. Patients will receive bendamustine at a total dose of 400mg/m2, divided in two doses of 200mg/m2/day on days -4 and -3. Melphalan is given at a total dose of 200mg/m2, divided in two doses of 100mg/m2/day, each on days -2 and -1, with the ASCT at day 0.
  Other Names: Ribomustin
  Arms: Arm B (BenMel)

SUMMARY:
Two high-dose chemotherapy regimens (melphalan alone versus the combination of melphalan and bendamustine) used for conditioning treatment before autologous stem cell transplantation will be compared in a 1:1 randomization in myeloma patients. The experimental arm is the bendamustine and melphalan (BenMel) combined regimen. The melphalan alone (Mel) regimen is the control (standard) treatment. Despite remarkable progress using novel agents both for induction before ASCT as well for maintenance after ASCT, definite cure in myeloma patients remains exceptional due to residual disease escaping intensive treatment. The aim of the study is to show an improvement of the rate of complete Remission 60 days after ASCT in myeloma patients from 50% with melphalan alone to 65% with the combination of bendamustine and melphalan.

DETAILED DESCRIPTION:
Background and Rationale:

High-dose chemotherapy with melphalan and autologous stem cell transplantation (ASCT) remains an integral component of the myeloma treatment algorithm for patients considered eligible for the procedure, nowadays performed in myeloma patients up to the age of 75 years. Despite remarkable progress using novel agents both for induction before ASCT as well for maintenance after ASCT, definite cure in myeloma patients remains exceptional due to residual disease escaping intensive treatment. Martino et al. recently reported data on the feasibility and efficacy of the combination of bendamustine and melphalan (BenMel) as a conditioning regimen to second ASCT in patients with myeloma. In addition, extensive experience is available on the use of bendamustine (200mg/m2/day given on days -7 and -6) together with melphalan (140mg/m2/day day -1) and two additional drugs, cytarabine and etoposide (each on days -5 to -2) in the BeEAM conditioning regimen which is increasingly used as the standard conditioning regimen in lymphoma patients, also in the investigators' clinic, with an acceptable tolerability and safety profile. In summary, these data suggest that combinations of melphalan and bendamustine are usually well tolerated and that the maximum tolerated dose of bendamustine is not reached with the doses of 200mg/m2/day given on two days added to melphalan,etoposide and cytarabine (BeEAM regimen). The investigators therefore suggest in this study to directly compare bendamustine 200 mg/m2/day (on days -4 and -3) plus melphalan 100mg/m2/day (on days -2 and -1) with melphalan 100mg/m2/day (days -2 and -1) in a randomized trial.

Objectives:

Primary objective To show a clinically meaningful improvement by 15% of the rate of complete remission (CR1) 60 days after ASCT in myeloma patients from 50% with melphalan alone to 65% with the combination of bendamustine and melphalan.

Secondary objectives To assess acute and late toxicities/adverse events (CTCAE 4.0) during the study period in patients treated with the combination of bendamustine and melphalan as compared to melphalan alone.

To assess the hematologic engraftment in patients treated with the combination of bendamustine and melphalan as compared to melphalan alone.

To particularly assess early renal toxicity in patients treated with the combination of bendamustine and melphalan as compared to melphalan alone.

To assess differences in overall survival and progression free survival in patients treated with the combination of bendamustine and melphalan as compared to melphalan alone after one year.

To assess the quality of life prior to ASCT and at day 60 assessment thereafter

Outcome:

To assess the rate of complete remission (CR1) 60 days after ASCT in myeloma patients treated with the combination of bendamustine and melphalan as compared to melphalan alone by routine laboratory myeloma parameters (serum M-gradient and light chain ratio) and bone marrow assessments in patients with CR1.

Number of Participants with Rationale: Applying a statistical power of 80% and a one-sided significance level of 20%, 60 evaluable patients will be needed in each group to show a clinically meaningful improvement by 15% of the rate of complete remission (CR1) 60 days after ASCT in myeloma patients, from 50% with melphalan alone to 65% with the combination of bendamustine and melphalan.

Study Duration: The total study duration is 36 months. Study design: Randomized two-arm open-label prospective phase II trial. Monitoring will be performed by the Clinical Trial Unit (CTU) of the University of Berne, Switzerland.

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP as well as all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Myeloma patients after standard first-line induction treatment. A second induction regimen in refractory myeloma patients is allowed.
* Patients must be considered being fit for subsequent consolidation with high-dose chemotherapy with melphalan with autologous stem cell support.
* Patients must be aged 18-75 years.
* Patients must have an ECOG < 3.
* Patients must have a creatinine clearance ≥ 40 ml/min.
* Patients must have a LVEF ≥ 40% within three months prior to start of study medication (Echo can be postponed to study treatment visit if clinically indicated).
* Female patients of child-bearing potential: No known pregnancy (a pregnancy test in female patients of child-bearing potential is not mandatory since patients are already under induction chemotherapy or mobilization chemotherapy, and pregnancy was excluded before starting chemotherapy…)
* Patients must have given voluntary written informed consent.

Exclusion Criteria:

* Patients with uncontrolled acute infection.
* Patients with a transplantation comorbidity index (HCTCI) > 6 points.
* Patients with concurrent malignant disease with the exception of basalioma/spinalioma of the skin or early-stage cervix carcinoma, or early-stage prostate cancer. Previous treatment for other malignancies (not listed above) must have been terminated at least 24 months before registration and no evidence of active disease shall be documented since then.
* Patients with major coagulopathy or bleeding disorder.
* Patients with other serious medical condition that could potentially interfere with the completion of treatment according to this protocol or that would impair tolerance to therapy or prolong hematological recovery.
* Lack of patient cooperation to allow study treatment as outlined in this protocol.
* Pregnancy or lactating female patients.
* The use of any anti-cancer investigational agents within 14 days prior to the expected start of trial treatment.
* Contraindications and hypersensitivity to any of the active chemotherapy compounds.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pabst, MD, Study Chair — Department of Medical Oncology, University Hospital Bern
Locations (1):
- Department for Medical Oncology University Hospital/Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Mel) | Arm B (BenMel)
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Mel) | Arm B (BenMel) | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 29 | 65
  >=65 years | 24 | 31 | 55
Age, Continuous [Median (Full Range); unit: years] | 62 [35 to 74] | 65 [46 to 74] | 63 [35 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 44
  Male | 35 | 41 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate
Description: Number of Patient achieving complete remissions (CR1) at 60 days after ASCT
Time Frame: 60 days
Population: Response rates were assessed according to the International Myeloma Working Group (IMWG). Bone marrow (BM) was assessed by cytomorphology, histopathology with immunohistochemistry, and immunophenotyping by multiparameter flow cytometry (MFC) for detection of measurable residual disease (MRD). MRD negativity was defined by less than 10-5 aberrant plasma cells after measuring at least 1000000 nucleated cells.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Mel) | Arm B (BenMel)
Number analyzed (Participants) | 60 | 60
Participants | 31 | 42

2. Secondary Outcome: Adverse Events
Description: Number of Patient experiencing toxicities/adverse events assessed according to the CTCAE 4.0 during the study period
Time Frame: 60 days
Population: Clinical assessment and documentation of toxicities exceeding grade II during hospitalization were performed until 60 days after ASCT.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Mel) | Arm B (BenMel)
Number analyzed (Participants) | 60 | 60
Participants | 36 | 43

3. Secondary Outcome: Hematologic Engraftment After High-dose Chemotherapy
Description: Number of days needed to achieve hematologic engraftment after high-dose chemotherapy induced myelosuppression is defined as the first day of neutrophils rising again above 0.5 G/l, and of platelets rising again above 20 G/L in the absence of platelet transfusions in the previous 3 days.
Time Frame: 30 days
Population: Time to neutrophil engraftment was defined as the duration between day 0 and the first 3 days of neutrophils >0.5 × 109/L after ASCT.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm A (Mel) | Arm B (BenMel)
Number analyzed (Participants) | 60 | 60
days | 12 [10 to 18] | 11 [10 to 60]

4. Secondary Outcome: Overall Survival
Description: Overall survival - Percentage of Participants Alive at 12 Months
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Mel) | Arm B (BenMel)
Number analyzed (Participants) | 60 | 60
percentage of participants | 96 | 96

5. Secondary Outcome: Quality of Life: EORTC Q30 Questionnaire
Description: Assessment of quality of life prior to ASCT and 60 days thereafter. The EORTC Q30 questionnaire will be given to patients at screening and at the day 60 assessment.
Time Frame: 60 days
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: Deaths were assessed up to 24 months. Adverse Events were assessed through 60 days
Arm/Group | Arm A (Mel) | Arm B (BenMel)
All-Cause Mortality (participants affected / at risk) | 0/60 | 1/60
Serious Adverse Events (participants affected / at risk) | 9/60 | 12/60
Other Adverse Events (participants affected / at risk) | 36/60 | 43/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Mel) (N=60) | Arm B (BenMel) (N=60)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
fever unkown origin (Infections and infestations) | 1 (1) | 0 (0)
neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
weakness (General disorders) | 1 (1) | 0 (0)
respiratory failue (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
fever (General disorders) | 0 (0) | 1 (1)
renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
right ventricular disfunction (Cardiac disorders) | 0 (0) | 1 (1)
weakness (General disorders) | 0 (0) | 1 (1)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Pancolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
weight loss (General disorders) | 0 (0) | 1 (1)
Panaritium (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Septic Schock (Infections and infestations) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Mel) (N=60) | Arm B (BenMel) (N=60)
Gastrointestinal disordes (Gastrointestinal disorders) | 31 (31) | 30 (30)
Metabolic and nutritional disorders (Metabolism and nutrition disorders) | 10 (10) | 20 (20)
Cardiac and thromboembolic disorders (Cardiac disorders) | 5 (5) | 3 (3)
Weight loss >10% (General disorders) | 0 (0) | 5 (5)
Engraftment syndrome (General disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT03187223/Prot_SAP_000.pdf